CLINICAL TRIAL: NCT05229757
Title: The Effect of Family Education on Functional Level, Activity Level and Families in Children With Cerebral Palsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Mehmet Ergun Kayiran, Msc, PT, Hasan Kalyoncu University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021/048
Record Dates: First submitted 2022-01-13; First posted 2022-02-08 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-02

CONDITIONS: Children With Cerebral Palsy
MeSH Terms: interventions — Physical Therapy Modalities; Rehabilitation; Rehabilitation Centers

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: The individuals included in the study and their families were not informed about which group they belonged to.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental): Children with cerebral palsy in the patient group received treatment in a special education and rehabilitation center two days a week for 8 weeks.
  Interventions: Other: Physiotherapy and rehabilitation treatment in a special education and rehabilitation center.
- Control Group (Active Comparator): Individuals in the control group were followed with a home program for 8 weeks.
  Interventions: Other: Family-based home exercise.

INTERVENTIONS:
Other: Physiotherapy and rehabilitation treatment in a special education and rehabilitation center. — Routine physiotherapy and rehabilitation practice was performed 2 days a week for 8 weeks in the special education and rehabilitation center.
  Arms: Study Group
Other: Family-based home exercise. — Home exercise was applied by the families every day of the week for 8 weeks.
  Arms: Control Group

SUMMARY:
The activity status of children with cerebral palsy between the ages of 3 and 18 who participated in the physiotherapy program in special education institutions throughout the province of Gaziantep was evaluated. The effect of the family education to be given on the activity status of the children and the psychosocial status of the families was investigated.

The individuals included in the study were divided into two groups as patient and control. In the beginning, the scales used to determine the activity status and the scales to determine the depression status of their families were applied in order to determine the status of both groups. Children with cerebral palsy in the patient group received treatment in a special education and rehabilitation center two days a week for 8 weeks. Individuals in the control group were followed up with a home program. After 8 weeks of treatment, the same tests were repeated and it was examined whether the family education provided made a difference in children with cerebral palsy and their parents.

ELIGIBILITY:
Inclusion Criteria:

* Be in the age range of 3-18 years.
* Getting a diagnosis of cerebral palsy.
* Agree to participate in the study.

Exclusion Criteria:

* If the child interrupts supportive education for any reason,
* Failure of the family to ensure continuity in participation

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 28 (Actual)
Dates: Start 2021-05-19 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
Abilhand Kids (For patients) | Change from Baseline Abilhand Kids at 8 weeks.
  It is a questionnaire consisting of 21 questions designed to test children's manual abilities. The applicability of the items by the child is evaluated in 3 steps as impossible, easy and difficult.
GMFM 66 (For patients) | Change from Baseline GMFM 66 at 8 weeks.
  Gross motor function assessment is a computerized test consisting of 66 questions. Evaluates the sub-titles as Reaching-Rolling, Sitting, Standing and running-Jumping.
PEDI (For patients) | Change from Baseline PEDI at 8 weeks.
  It is a scale that evaluates the functional skills of the child and the help and manner of the caregiver, in which each part is evaluated separately as self-care, mobility and social function items.
Beck Depression Scale (For family) | Change from Baseline Beck Depression Scale at 8 weeks.
  It is a survey aiming to reach the result by scoring between 0 and 3 with 21 questions. According to the total score, it is divided into 4 groups as minimal, mild, moderate and severe depression.
IPFAM (For family) | Change from Baseline IPFAM at 8 weeks.
  The family impact scale asks for answers in 4 categories: I strongly disagree (4 points), disagree (3 points), agree (2 points), completely agree (1 point) in 27 questions. Makes classification according to the total score.

CONTACTS AND LOCATIONS:
Locations (1):
- Hasan Kalyoncu University, Gaziantep, Şahinbey, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No